CLINICAL TRIAL: NCT06137898
Title: The Benefits of Dietary and Micro-nutritional Management for Well-being at Work
Acronym: MEDEIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Larena SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: PIL-RIPH3-MEDEIS-023
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: biological check-up — Blood sampling

SUMMARY:
The aim of this observational study is to describe the benefits of this treatment, particularly in terms of changes in the well-being of participating employees in relation to their nutritional/micro-nutritional status.

DETAILED DESCRIPTION:
Biological check-ups and medical appointments with the investigators will be carried out as part of the hygienic-dietary and micro-nutritional management that study participants have enrolled in. No additional investigations or blood sampling are required for the study. Participants will only be asked to complete the WHO5 and MSP9 self-questionnaires once a month, for 12 months. The inclusion visit will take place at the same time as the first medical visit for dietary and nutritional management. After obtaining the participant's non-opposition, the investigator will check the inclusion and non-inclusion criteria.

If eligible, the participant will download a data collection application onto his or her smartphone, and will be provided with an identifier and access code.

As part of the program, dietary hygiene and micro-nutritional recommendations will be proposed on the basis of the results of a biological (blood test) and nutritional (interview with the doctor) assessment. If necessary, the doctor may prescribe additional blood tests on a regular basis, and will carry out nutritional assessments to adapt the program's management.

The program will be organized into 5 visits:

* a first visit V0 (micro-nutritional interview) with a biological check-up ;
* a second V1 visit (within a fortnight of the initial visit) to review all the results of the initial assessment and, if necessary, to implement hygienic-dietary and/or nutritional recommendations (in the form of cards) and/or a micro-nutritional prescription;
* quarterly follow-up visits (at 3 and 6 months) and a visit at 1 year to carry out check-ups.

These visits can take place face-to-face with an investigating physician, or by teleconsultation.

A statistical analysis plan will precisely indicate the populations studied, the analysis procedures, the treatment of missing data envisaged, the statistical tests for each variable and for the analysis of the primary and secondary judgment criteria to be used.

The threshold of statistical significance will be defined at the risk alpha = 0.05.

Trial data will be collected :

* by investigators for biological and clinical data on the e-CRF
* by participants on their smartphones using the data acquisition system for self-questionnaires.

Description of the population:

Descriptions of subjects included in the study will be made by mean and standard deviation for quantitative variables and by frequency and numbers for qualitative variables.

Analysis of endpoints:

Changes in WHO5, MSP9 scores and biological variables will be analyzed using a repeated-measures ANOVA. The same analyses will be carried out on secondary criteria. Correlations between changes in WHO5 and MSP-9 scores and changes in biological and clinical and clinical data.

Sample size:

The required sample size is based on the evolution of the WHO-5 global score between the initial visit and the 6-month follow-up visit using a two-tailed paired t-test with an estimated mean evolution of 5, an estimated standard deviation of 19 (12) and a confidence level of 90. 154 subjects are required, which is rounded up to 200 to account for unexploitable records (≈10%) or premature study withdrawals (≈10%).

ELIGIBILITY:
Inclusion Criteria:

* Wishing to initiate dietetic and micro-nutritional management of their state of health
* Having freely declared to the investigator that he/she does not object to his/her participation in the study the study and to the collection of data strictly necessary for the study, after having received informed oral and written information from the investigator
* Have a smartphone compatible with the secure data collection application

Exclusion Criteria:

* Pregnant or breast-feeding women
* Participating in another study or in the exclusion period
* Person under court protection

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult wishing to initiate dietetic and micro-nutritional management of their state of health
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of WHO-5 | Baseline, 6 months
  Evolution of World Health Organization Well-Being Index score (WHO 5) between M0 inclusion (V1) and 6 months after the start of management (V3).

SECONDARY OUTCOMES:
Evolution of subjective well-being | Each month up to 12 months
  Evolution of the WHO-5 score between M0 inclusion (V1) and each month of management to M12
Evolution of psychological stress | Each month up to 12 months
  Evolution of psychological stress measured using the MSP9 scale between inclusion M0 (V1) and each month of treatment up to M12.
Evolution of biological parameters | Baseline, Month 3, Month 6, Month 12
  Evolution of biological parameters (nutritional/micro-nutritional status) measured at inclusion and at the visits usually organized as part of the management process. (M0, M3, M6, M12).
Prevention and evolution of symptomatologies mainly linked to nutritional nutritional/micro-nutritional status | Baseline, Month 3, Month 6, Month 12
  the micro-nutritional follow-up questionnaire completed at inclusion and at the usual follow-up visits (M0, M3, M6, M12).
Describe compliance with hygienodietary and micro-nutritional follow-up. | Baseline, Month 3, Month 6, Month 12
  Compliance will be described by an observance questionnaire completed at inclusion and at the usual follow-up visits (M0, M3, M6 and M12), and by attendance (presence/absence at the various follow-up follow-up visits).
Describe satisfaction with hygienodietary and micro-nutritional follow-up. | Month 3, Month 6, Month 12
  Satisfaction with care will be described using 4-point Likert scales (0: not at all satisfied to 3: very satisfied) completed at follow-up visits (M3, M6 and M12).

CONTACTS AND LOCATIONS:
Overall Officials: Carole PERRIN, Principal Investigator — CEN
Locations (1):
- CEN, Dijon, France